CLINICAL TRIAL: NCT07137182
Title: The Effect of Physical Activity on Cardiovascular Disease Risk Awareness and Self-Worth in Young Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Hatice YAĞCI KARAMANLI, Principal Investigator, Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 04-2025/57
Record Dates: First submitted 2025-08-07; First posted 2025-08-22 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular (CV) Risk; Physical Activities
Keywords: cardiovascular risk; physical activities; self worth
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The type of this study is a randomized controlled trial with a pre-test post-test model, including experimental and control groups.
Who Masked: Outcomes Assessor
Masking Description: The statistician who will perform the analyses will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deney (Experimental): group to be included in the application
  Interventions: Other: 8-week physical activity program
- kontrol (No Intervention): no intervention will be made

INTERVENTIONS:
Other: 8-week physical activity program — Individuals in the experimental group will be administered an eight-week physical activity program. The researcher who will administer the activity is a specialist in Sports Sciences and holds the necessary certifications. The activity program includes cardio exercises, jumping, stretching, and stretching exercises.
  Arms: Deney

SUMMARY:
The main purpose of this study was to reveal the self-worth perceptions of women who regularly participate in physical activity and to investigate the effect of physical activity on self-worth perception and cardiovascular risk awareness.

DETAILED DESCRIPTION:
International activity is one of the most important elements of maintaining a healthy life and contributes to the enhancement of life. According to the World Health Organization (WHO), physical activity is defined as any activity that involves the movement of body muscles and involves a certain amount of energy expenditure. Physical activity for university undergraduates includes a variety of movements, either individually or in groups. These activities include exercises performed in rotation or in open spaces, sports competitions, games that involve movement, running, jumping, and exercises performed in physical education classes.

Physical activity is important for many aspects of health. Despite this, participation in health-enhancing physical activities is quite low. Consequently, physical activity has become a serious public health issue today. It is known that women, in particular, participate less in physical activity than men. Participation in regular physical activity can improve women's health and prevent major causes of disease and death. The World Health Organization (WHO) has linked the reasons for women's physical inactivity to constraints such as lower income, family responsibilities, and cultural differences. Regular physical activity plays an important role in reducing the risk of diseases such as heart disease, type 2 diabetes, obesity, hypertension, and colon cancer.

In recent years, an increase in studies focusing on women's health and physical activity has been observed. Physical activity-focused research also focuses on the psychological and social impacts of women, such as quality of life, cognitive function, depression, leisure satisfaction, self-esteem, anthropometry, nutritional habits, balance-mobility, and eating behaviors. In addition to physical improvements, there are also studies in the field of health that reveal individuals' psychological and social well-being.

In addition to social situations, individuals' psychological perceptions of self-worth are seen as one of the most important factors determining their lives. The concept of self-worth is considered a key figure in psychological well-being and is seen as the key to happiness and success. Furthermore, self-worth encompasses a person's self-definition and evaluation, as well as their analysis of their own worth or individual worth. Perception of self-worth is a crucial factor in improving both mental and physical health.

Based on the information provided, the primary objective of this study is to explore the self-worth perceptions of women who regularly participate in physical activity and to investigate the impact of physical activity on self-worth perception and cardiovascular risk awareness.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* Voluntarily participating in the study
* Being female

Exclusion Criteria:

* Having any physical disability,
* Having had an injury or accident,
* Being pregnant or having recently given birth,
* Having a cognitive impairment that would prevent completing the survey and maintaining communication,

Min Age: 18 Weeks | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Kadın
Enrollment: 60 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-11-21 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Female Physical Active Self-Esteem Scale | 8 weeks
  The Women's Physical Activity Self-Esteem Scale, developed by Huberty et al. (22) and validated and validated in Turkish by Yurtçiçek Ergüntop and Kömürcü (23), was used to measure women's physical activity self-esteem. The scale's Cronbach's alpha (0.91) and split-half value (0.74) were above 0.70, indicating reliability. The scale consists of a total of 37 items.
Cardiovascular Disease Risk Awareness Assessment Scale | 8 weeks
  The 26-item shortened version of the scale was adapted by Woringer et al., and the Turkish validity and reliability study was conducted by Doğru et al. (24,25). The scale consists of three sub-dimensions (perceived heart attack/stroke risk, perceived benefits and intentions to change, and healthy eating intentions).

CONTACTS AND LOCATIONS:
Overall Officials: Hatice YAĞCI KARAMANLI, Principal Investigator — KARAMANOĞLU MEHMETBEY UNİVERSTY

IPD SHARING:
Plan to Share IPD: No
Consent to share data was not obtained from all co-authors.